CLINICAL TRIAL: NCT05703724
Title: Prevalence of Glaucoma in Belgium: a Multicenter National Trial
Acronym: BelGlaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Santen Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: S66402
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects (Other): A fundus picture will be acquired without pupil dilation. This examination will be followed by an intra-ocular pressure measurement. The results will be discussed with the participating subject by the present physician. For each subject, both eyes will be evaluated. In case of suspected glaucoma, the subject will be referred to an ophthalmologist for further evaluation.
  Interventions: Device: AI algorithm for the detection of glaucoma

INTERVENTIONS:
Device: AI algorithm for the detection of glaucoma — The investigational device that will be used during this study is an AI algorithm embedded into an API for the detection of glaucoma developed by MONA.health

SUMMARY:
To screen for the presence of glaucoma in a Belgian population over 40 years old using an AI algorithm developed for the detection of glaucoma based on fundus pictures.

DETAILED DESCRIPTION:
In this study, we aim to detect individuals with glaucoma and refer them for further evaluation and treatment when necessary. In so doing, we want to get an estimation of the prevalence of glaucoma in the Belgian population of 40+ years.

A fundus picture will be acquired without pupil dilation. This examination will be followed by an intra-ocular pressure measurement. The results will be discussed with the participating subject by the present physician. For each subject, both eyes will be evaluated. In case of suspected glaucoma, the subject will be referred to an ophthalmologist for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years or above

Exclusion Criteria:

* Aged under 40 years
* Insufficient knowledge of Dutch, French or English required to complete the imaging protocol and questionnaire
* Physical or mental inability to participate

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1418 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of glaucoma in Belgium | 4 months
  To study the prevalence of glaucoma in the Belgian population over 40 years old

SECONDARY OUTCOMES:
Validation of AI algorithm | 7 months
  To validate an existing AI-based algorithm for automatic detection of glaucoma

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven
Locations (8):
- Belgium (8):
  - UZA, Edegem, Antwerpen
  - Saint-Luc (UCL), Brussels, Brussels Capital
  - Hôpital Erasme, Brussels, Brussels Capital
  - CHU Liège, Liège, Luik
  - AZ Sint-Lucas, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - AZ Sint-Jan, Bruges, West-Vlaanderen
  - ZNA Middelheim, Antwerp

IPD SHARING:
Plan to Share IPD: No